CLINICAL TRIAL: NCT06128733
Title: A Phase I/II, Randomized, Descriptive, Safety and Immunogenicity Study to Assess Pentavalent Meningococcal ABCYW Vaccine Formulations in Adults (18 to 25 Years of Age) and Adolescents (10 to 17 Years of Age).
Brief Title: Study of an Investigational Pentavalent Meningococcal ABCYW Vaccine in Adults and Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAN00010; U1111-1272-6824 (Registry Identifier: ICTRP); 2023-000924-13 (EudraCT Number)
Record Dates: First submitted 2023-10-26; First posted 2023-11-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Meningococcal Immunisation; Healthy Volunteers
MeSH Terms: interventions — 4CMenB vaccine; MenB-FHbp vaccine; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Modified double-blind: in order to maintain the blind, a placebo injection will be given and blood sample will be collected from all participants at each visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1: MenPenta Formulation 1 (Experimental): Participants (ACWY naive and primed adults or adolescents) will receive injections of the pentavalent meningococcal ABCYW vaccine and placebo
  Interventions: Biological: Pentavalent Meningococcal ABCYW vaccine; Biological: Placebo
- Group 2: MenPenta Formulation 2 (Experimental): Participants (ACWY naive and primed adults or adolescents) will receive injections of the pentavalent meningococcal ABCYW vaccine and placebo
  Interventions: Biological: Pentavalent Meningococcal ABCYW vaccine; Biological: Placebo
- Group 3: Bexsero® + Menveo® (Active Comparator): Participants (ACWY naive and primed adults or adolescents) will receive injections of Bexsero® + Menveo® vaccine
  Interventions: Biological: Meningococcal group B vaccine; Biological: MenACYW conjugate vaccine
- Group 4: Trumenba® + Menveo® (Active Comparator): Participants (ACWY naive and primed adults or adolescents) will receive injections of Trumenba® + Menveo® vaccine
  Interventions: Biological: Meningococcal group B vaccine; Biological: MenACYW conjugate vaccine
- Group 5: MenQuadfi® (Active Comparator): Participants (ACWY naive and primed adults or adolescents) will receive injections of MenQuadfi® vaccine and placebo
  Interventions: Biological: MenACYW conjugate vaccine; Biological: Placebo
- Group 6: Sanofi MenB (Experimental): Participants (ACWY naive and primed adults or adolescents) will receive injections of SP MenB vaccine and placebo
  Interventions: Biological: Meningococcal group B vaccine; Biological: Placebo
- Group 7: PENBRAYA (Active Comparator): Participants (ACWY naive and primed adolescents) will receive injections of PENBRAYA vaccine and placebo
  Interventions: Biological: MenABCYW conjugate vaccine

INTERVENTIONS:
Biological: Pentavalent Meningococcal ABCYW vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular (IM)
  Other Names: MenPenta
  Arms: Group 1: MenPenta Formulation 1; Group 2: MenPenta Formulation 2
Biological: MenACYW conjugate vaccine — Pharmaceutical form:Solution for injection in vial-Route of administration:Intramuscular (IM)
  Other Names: MenQuadFi®
  Arms: Group 5: MenQuadfi®
Biological: Meningococcal group B vaccine — Pharmaceutical form:Suspension for injection in pre-filled syringe-Route of administration:Intramuscular (IM)
  Other Names: Bexsero®
  Arms: Group 3: Bexsero® + Menveo®
Biological: Meningococcal group B vaccine — Pharmaceutical form:Suspension for injection in pre-filled syringe-Route of administration:Intramuscular (IM)
  Other Names: Trumenba®
  Arms: Group 4: Trumenba® + Menveo®
Biological: Meningococcal group B vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular (IM)
  Other Names: Sanofi MenB
  Arms: Group 6: Sanofi MenB
Biological: MenACYW conjugate vaccine — Pharmaceutical form:Powder and solvent for solution for injection-Route of administration:Intramuscular (IM)
  Other Names: Menveo®
  Arms: Group 3: Bexsero® + Menveo®; Group 4: Trumenba® + Menveo®
Biological: Placebo — Pharmaceutical form:Solution for injection in vial-Route of administration:Intramuscular (IM)
  Arms: Group 1: MenPenta Formulation 1; Group 2: MenPenta Formulation 2; Group 5: MenQuadfi®; Group 6: Sanofi MenB
Biological: MenABCYW conjugate vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular (IM)
  Other Names: PENBRAYATM
  Arms: Group 7: PENBRAYA

SUMMARY:
The purpose of VAN00010 study is to assess the safety and immunogenicity of the investigational pentavalent meningococcal ABCYW vaccine in adults and adolescents.

The study duration will be up to 12 months for all participants.

DETAILED DESCRIPTION:
The study duration will be approximately 12 months for all participants

ELIGIBILITY:
Inclusion Criteria: - Aged 18 to 25 years or 10 to 17 years on the day of inclusion

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and judgment of the Investigator.
* Participants who are either unvaccinated with MenACWY vaccine or have received a single previous dose of MenACWY vaccine at least 4 years prior to study enrollment Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:
* Known or suspected congenital or acquired immunodeficiency
* History of any Neisseria meningitidis infection
* At high risk for meningococcal infection during the study
* Individuals with active tuberculosis
* History of Guillain-Barré syndrome
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion NOTE: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1215 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events (AEs) | Within 30 minutes after each vaccination
  Unsolicited systemic AEs that occur within 30 minutes after vaccination
Number of participants with solicited injection site reactions or systemic reactions | Within 7 days after each vaccination
  Pre-defined solicited injection site reactions and systemic reactions that are pre-listed in the diary cards and CRF
Number of participants with unsolicited AEs | Within 30 days after each vaccination
  Non-serious AEs other than solicited reactions
Number of participants with serious adverse events (SAEs) | From baseline up to 12 months
  SAEs (including adverse events of special interest [AESIs]) reported throughout the study
Number of participants with medically attended adverse events (MAAEs) | From baseline up to 12 months
  An MAAE is a new onset or a worsening of a condition that prompts the participant or participant's parent/legally acceptable representative to seek unplanned medical advice at a physician's office or Emergency Department
Number of participants with out-of-range biological test results | Before each vaccination up to 7 days after primary vaccination visits in the sentinel cohorts (the first 5 participants enrolled in each vaccine group) of each age group
hSBA meningococcal serogroups A, C, W, and Y vaccine seroresponse pre-dose and 1 month after the second dose in adolescent participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 7)
  Seroresponse defined as post-second vaccination titers ≥ 1:16 for participants with pre-vaccination hSBA titers < 1:4 or post-second vaccination titers ≥ 4 times the pre-vaccination titer for participants with a pre-vaccination titer more than or equal to the lower limit of quantification (LLOQ)
hSBA meningococcal serogroups A, C, W, and Y antibody titers pre-dose and 1 month after the second dose in adolescent participants | Day 211 (for Group 1 to 7)
  hSBA titers ≥ 1:8
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroups A, C, W and Y pre-dose and 1 month after the second dose in adolescent participants | Day 01 (pre-dose) and Day 31 Day 211 (for Group 1 to 7)
  Geometric mean titers
Percentage of participants with hSBA titers more or equal to lower limit of quantification (LLOQ) against each of serogroups A, C, W, and Y in adolescent participants | Day 01 (pre-dose) Day 211 (for Group 1 to 7)
hSBA meningococcal serogroup B seroresponse pre-dose and 1 month after second dose in adolescent participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 7)
  Seroresponse defined as a 4-fold increase in hSBA titers
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference MenB strains) ≥ 1:4 pre-dose 1 and 1 month post-second dose in adolescent participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 7)
  hSBA titers ≥ 1:4 for reference MenB strains
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference MenB strains) ≥ 1:8 pre-dose 1 and 1 month post-second dose in adolescent participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 7)
  hSBA titers ≥ 1:8 for reference MenB strains
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroup B (reference MenB strains) pre-dose 1 and 1 month post-second dose in adolescent participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 7)
  Geometric mean titers for the reference MenB strains
Percentage of participants with hSBA titers more or equal to lower limit of quantification (LLOQ) against each and all serogroups B (reference MenB strains) in adolescent participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 7)

SECONDARY OUTCOMES:
hSBA meningococcal serogroups A, C, W, and Y vaccine seroresponse at each timepoint | D01 (pre-dose) and D31 (post-dose 1 and pre-dose 2), D61 (post-dose 2), D181 (pre-dose 3) and D211 (post-dose 3) for adults (Group 1-6). D01 (pre-dose) and D31 (post-dose 1), D181 (pre-dose 2) and D211 (post-dose 2) for adolescents (Group 1-7)
  Seroresponse defined as post-vaccination titers ≥ 1:16 for participants with pre-vaccination titers < 1:4 or post-vaccination titer ≥ 4 times the pre-vaccination titer for participants with pre-dose 1 vaccination titers more than the lower limit of quantification (LLOQ)
hSBA meningococcal serogroups A, C, W, and Y antibody titers at each timepoint | D01 (pre-dose) and D31 (post-dose 1 and pre-dose 2), D61 (post-dose 2), D181 (pre-dose 3) and D211 (post-dose 3) for adults (Group 1-6). D01 (pre-dose) and D31 (post-dose 1), D181 (pre-dose 2) and D211 (post-dose 2) for adolescents (Group 1-7)
  hSBA titers ≥ 1:8 post-vaccination
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroups A, C, W and Y at each timepoint | D01 (pre-dose) and D31 (post-dose 1 and pre-dose 2), D61 (post-dose 2), D181 (pre-dose 3) and D211 (post-dose 3) for adults (Group 1-6). D01 (pre-dose) and D31 (post-dose 1), D181 (pre-dose 2) and D211 (post-dose 2) for adolescents (Group 1-7)
  Geometric mean titers
Percentage of participants with hSBA titers more or equal to LLOQ against each of serogroups A, C, W, and Y at each timepoint | D01 (pre-dose) and D31 (post-dose 1 and pre-dose 2), D61 (post-dose 2), D181 (pre-dose 3) and D211 (post-dose 3) for adults (Group 1-6). D01 (pre-dose) and D31 (post-dose 1), D181 (pre-dose 2) and D211 (post-dose 2) for adolescents (Group 1-7)
hSBA meningococcal serogroup B (reference MenB strains) vaccine seroresponse at each timepoint | D01 (pre-dose) and D31 (post-dose 1 and pre-dose 2), D61 (post-dose 2), D181 (pre-dose 3) and D211 (post-dose 3) for adults (Group 1-6). D01 (pre-dose) and D31 (post-dose 1), D181 (pre-dose 2) and D211 (post-dose 2) for adolescents (Group 1-7)
  Seroresponse defined as a 4-fold increase in hSBA titers
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference MenB strains) ≥ 1:4 at each timepoint | D01 (pre-dose) and D31 (post-dose 1 and pre-dose 2), D61 (post-dose 2), D181 (pre-dose 3) and D211 (post-dose 3) for adults (Group 1-6). D01 (pre-dose) and D31 (post-dose 1), D181 (pre-dose 2) and D211 (post-dose 2) for adolescents (Group 1-7)
  hSBA titers ≥ 1:4 for reference MenB strains
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference MenB strains) ≥ 1:8 at each timepoint | D01 (pre-dose) and D31 (post-dose 1 and pre-dose 2), D61 (post-dose 2), D181 (pre-dose 3) and D211 (post-dose 3) for adults (Group 1-6). D01 (pre-dose) and D31 (post-dose 1), D181 (pre-dose 2) and D211 (post-dose 2) for adolescents (Group 1-7)
  hSBA titers ≥ 1:8 reference MenB strains
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroup B (reference MenB strains) at each timepoint | D01 (pre-dose) and D31 (post-dose 1 and pre-dose 2), D61 (post-dose 2), D181 (pre-dose 3) and D211 (post-dose 3) for adults (Group 1-6). D01 (pre-dose) and D31 (post-dose 1), D181 (pre-dose 2) and D211 (post-dose 2) for adolescents (Group 1-7)
  Geometric mean titers for reference MenB strains
Percentage of participants with hSBA composite seroresponse titers more or equal to LLOQ for reference MenB strains for each timepoint | D01 (pre-dose) and D31 (post-dose 1 and pre-dose 2), D61 (post-dose 2), D181 (pre-dose 3) and D211 (post-dose 3) for adults (Group 1-6). D01 (pre-dose) and D31 (post-dose 1), D181 (pre-dose 2) and D211 (post-dose 2) for adolescents (Group 1-7)
hSBA meningococcal serogroup B (reference and additional MenB strains) vaccine seroresponse pre-dose 1 and 1 month post-second and third dose in adolescent participants | Day 01 (pre-dose), Day 61 (post-dose 2) and Day 211 (post-dose 3) (for Group 1 to 6 for adults) and Day 211 (for Group 1 to 7 for adolescents)
  Seroresponse defined as a 4-fold increase in hSBA titers from D01 to post-vaccination for reference and additional MenB strains
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference and additional MenB strains) ≥ 1:4 pre-dose 1 and 1 month post-second and third dose in adolescent participants | Day 01 (pre-dose), Day 61 (post-dose 2) and Day 211 (post-dose 3) (for Group 1 to 6 for adults) and Day 211 (for Group 1 to 7 for adolescents)
  hSBA titers ≥ 1:4 for reference and additional MenB strains
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference and additional MenB strains) ≥ 1:8 pre-dose 1 and 1 month post-second and third dose in adolescent participants | Day 01 (pre-dose), Day 61 (post-dose 2) and Day 211 (post-dose 3) (for Group 1 to 6 for adults) and Day 211 (for Group 1 to 7 for adolescents)
  hSBA titers ≥ 1:8 for reference and additional MenB strains
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroup B (reference and additional MenB strains) pre-dose 1 and 1 month post-second and third dose in adolescent participants | Day 01 (pre-dose), Day 61 (post-dose 2) and Day 211 (post-dose 3) (for Group 1 to 6 for adults) and Day 211 (for Group 1 to 7 for adolescents)
  Geometric mean titers for reference and additional MenB strains
Percentage of participants with hSBA composite seroresponse titers more or equal to LLOQ reference and additional MenB strains in adolescent participants | Day 01 (pre-dose), Day 61 (post-dose 2) and Day 211 (post-dose 3) (for Group 1 to 6 for adults) and Day 211 (for Group 1 to 7 for adolescents)
hSBA meningococcal serogroups A, C, W, and Y vaccine seroresponse 1 month after the third dose in adult participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 6)
  Seroresponse defined as post-third vaccination titers ≥ 1:16 for participants with pre-vaccination hSBA titers < 1:4 or post-third vaccination titers ≥ 4 times the pre-vaccination titer for participants with a pre-vaccination titer more than the lower limit of quantification (LLOQ)
hSBA meningococcal serogroups A, C, W, and Y antibody titers pre-dose and 1 month after the third dose in adult participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 6)
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroups A, C, W and Y pre-dose and 1 month after the third dose in adult participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 6)
Percentage of participants with hSBA titers more or equal to LLOQ against each of serogroups A, C, W, and Y in adult participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 6)
hSBA meningococcal serogroup B (reference MenB strains) seroresponse pre-dose and 1 month after third dose in adult participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 6)
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference MenB strains) ≥ 1:4 pre-dose 1 and 1 month post-third dose in adult participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 6)
Percentage of Participants With Meningococcal Antibody Titers against meningococcal serogroup B (reference MenB strains) ≥ 1:8 pre-dose 1 and 1 month post-third dose in adult participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 6)
Geometric mean titers (GMTs) of Antibodies against Meningococcal Serogroup B (reference MenB strains) pre-dose 1 and 1 month post-third dose in adult participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 6)
Percentage of participants with hSBA titers more or equal to lower limit of quantification (LLOQ) against each and all serogroups B (reference MenB strains) in adult participants | Day 01 (pre-dose) and Day 211 (for Group 1 to 6)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (47):
- United States (46):
  - Accel Research Site - Birmingham Clinical Research Unit- Site Number : 8400080, Birmingham, Alabama
  - Lakeview Clinical Research Site Number : 8400029, Guntersville, Alabama
  - Alliance for Multispecialty Research- Phoenix- Site Number : 8400056, Tempe, Arizona
  - Harrisburg Family Medical Center Site Number : 8400070, Harrisburg, Arkansas
  - Smart Cures Clinical Research Site Number : 8400072, Anaheim, California
  - Hope Clinical Research, LLC- Site Number : 8400001, Canoga Park, California
  - Apex Research Group Site Number : 8400071, Fair Oaks, California
  - Velocity Clinical Research-Washington DC Site Number : 8400102, Washington D.C., District of Columbia
  - Accel Clinical Research-Deland Clinical Research Unit- Site Number : 8400081, DeLand, Florida
  - SIMEDHealth, LLC- Site Number : 8400045, Gainesville, Florida
  - Accel Research Sites-St. Petersburg-Largo- Site Number : 8400082, Largo, Florida
  - South Florida Research Organization Site Number : 8400086, Medley, Florida
  - Life Arc Research-Miami Site Number : 8400094, Miami, Florida
  - Charisma Medical and Research center Site Number : 8400097, Miami Lakes, Florida
  - Accel Research - Nona Pediatric Center Site Number : 8400079, Orlando, Florida
  - Ormond Beach Clinical Research- Site Number : 8400073, Ormond Beach, Florida
  - Palm Harbor Dermatology- Site Number : 8400030, Tampa, Florida
  - PAS Research Site Number : 8400032, Tampa, Florida
  - VICIS Clinical Research-Tampa Site Number : 8400065, Tampa, Florida
  - Leavitt Clinical Research-Idaho Falls- Site Number : 8400075, Idaho Falls, Idaho
  - Snake River Research, PLLC- Site Number : 8400100, Idaho Falls, Idaho
  - AES Peoria- Site Number : 8400090, Peoria, Illinois
  - AMR Evansville Site Number : 8400062, Evansville, Indiana
  - AMR - Newton- Site Number : 8400104, Newton, Kansas
  - ~Kentucky Pediatics / Adult Research- Site Number : 8400009, Bardstown, Kentucky
  - Michael W. Simon, MD, PSC- Site Number : 8400026, Lexington, Kentucky
  - Vida Clinical Studies Site Number : 8400084, Dearborn Heights, Michigan
  - Vida Clinical Studies- Site Number : 8400084, Dearborn Heights, Michigan
  - Be Well Clinical Studies- Site Number : 8400077, Lincoln, Nebraska
  - Alivation Research (Primary Care) Site Number : 8400046, Lincoln, Nebraska
  - Quality Clinical Research, Inc.- Site Number : 8400074, Omaha, Nebraska
  - Velocity Clinical Research, Omaha- Site Number : 8400066, Omaha, Nebraska
  - Velocity Clinical Research-Albuquerque- Site Number : 8400101, Albuquerque, New Mexico
  - Prime Global Research, Inc. Site Number : 8400043, The Bronx, New York
  - Monroe Biomedical Research - Site Number : 8400099, Monroe, North Carolina
  - SPICA Clinical Research Site Number : 8400098, Columbia, South Carolina
  - Coastal Carolina Research Center - N Charleston- Site Number : 8400050, North Charleston, South Carolina
  - Tribe Clinical Research at Parkside Pediatrics-Five Forks Site Number : 8400049, Simpsonville, South Carolina
  - Pediatric Clinical Trials Tullahoma- Site Number : 8400020, Tullahoma, Tennessee
  - New Horizon Medical Group-Houston Site Number : 8400069, Houston, Texas
  - DM Clinical Research- Bellaire- Site Number : 8400052, Houston, Texas
  - Advances in Health- Pearland- Site Number : 8400078, Pearland, Texas
  - Be Well Clinical Studies -Round Rock Site Number : 8400053, Round Rock, Texas
  - Progressive Clinical Research- Site Number : 8400028, Bountiful, Utah
  - AMR Utah-Wee Care Pediatrics-Kaysville- Site Number : 8400106, Kaysville, Utah
  - Alliance for Multispecialty Research- Site Number : 8400107, Murray, Utah
- Investigational Site Number : 6300001, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAN00010 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25521&tenant=MT_SNY_9011